CLINICAL TRIAL: NCT06999148
Title: Study on The Sensitizing Effect of Sonodynamic Therapy on The Treatment of Brainstem Glioma With Radiotherapy and Chemotherapy and Survival Analysis
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Yingjuan Zheng (Other)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other); Peking University (Other)
Responsible Party: Sponsor-Investigator, Yingjuan Zheng, Chief physician, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YZheng
Record Dates: First submitted 2025-05-11; First posted 2025-05-31 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Glioma (Any Grade) in the Brain
Keywords: Sonodynamic; Brainstem Gliomas; Radiotherapy; Chemotherapy
MeSH Terms: conditions — Glioma | interventions — Radiotherapy; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sonodynamictherapy (Experimental): SDT: Hematoporphyrin 5 mg/kg.Sonodynamic therapy is administered 40 hours later, twice a day with an interval of 10-12 hours, for 5 consecutive days. One cycle lasts 28 days, and a total of 4-6 cycles are conducted Radiotherapy: The dose is 50-54 Gy, 1.8-2 Gy per day, 5 times a week, for a total of 25 sessions Chemotherapy: When temozolomide is administered concurrently with radiotherapy, the dose is 75 mg/m² per day, taken daily until the end of radiotherapy. For adjuvant chemotherapy with temozolomide, the dose is 150 mg/m² per day from day1to day 5, followed by a 23-day rest period. Each cycle lasts 28 days. If well-tolerated, the dose should be adjusted to 200 mg/m² per day for the 2nd - 6th cycles Targeted Therapy: Bevacizumab 7.5-10 mg/kg, once every 3 weeks, for a total of 4-6 courses
  Interventions: Procedure: Sonodynamictherapy
- Control Group (Active Comparator): Radiotherapy: The dose is 50-54 Gy, 1.8-2 Gy per day, 5 times a week, for a total of 25 sessions Chemotherapy: When temozolomide is administered concurrently with radiotherapy, the dose is 75 mg/m² per day, taken daily until the end of radiotherapy. For adjuvant chemotherapy with temozolomide, the dose is 150 mg/m² per day from day 1 to day 5, followed by a 23 - day rest period. Each cycle lasts 28 days. If well - tolerated, the dose should be adjusted to 200 mg/m² per day for the 2nd - 6th cycles Targeted Therapy: Bevacizumab 7.5-10 mg/kg, once every 3 weeks, for a total of 4-6 courses
  Interventions: Drug: Radiotherapy plus temozolomide

INTERVENTIONS:
Procedure: Sonodynamictherapy — SDT: Hematoporphyrin 5 mg/kg.Sonodynamic therapy is administered 40 hours later, twice a day with an interval of 10-12 hours, for 5 consecutive days. One cycle lasts 28 days, and a total of 4-6 cycles are conducted Radiotherapy: The dose is 50-54 Gy, 1.8-2 Gy per day, 5 times a week, for a total of 25 sessions Chemotherapy: When temozolomide is administered concurrently with radiotherapy, the dose is 75 mg/m² per day, taken daily until the end of radiotherapy. For adjuvant chemotherapy with temozolomide, the dose is 150 mg/m² per day from day1to day 5, followed by a 23-day rest period. Each cycle lasts 28 days. If well-tolerated, the dose should be adjusted to 200 mg/m² per day for the 2nd - 6th cycles Targeted Therapy: Bevacizumab 7.5-10 mg/kg, once every 3 weeks, for a total of 4-6 courses
  Arms: Sonodynamictherapy
Drug: Radiotherapy plus temozolomide — Radiotherapy: The dose is 50-54 Gy, 1.8-2 Gy per day, 5 times a week, for a total of 25 sessions Chemotherapy: When temozolomide is administered concurrently with radiotherapy, the dose is 75 mg/m² per day, taken daily until the end of radiotherapy. For adjuvant chemotherapy with temozolomide, the dose is 150 mg/m² per day from day 1 to day 5, followed by a 23 - day rest period. Each cycle lasts 28 days. If well - tolerated, the dose should be adjusted to 200 mg/m² per day for the 2nd - 6th cycles Targeted Therapy: Bevacizumab 7.5-10 mg/kg, once every 3 weeks, for a total of 4-6 courses
  Arms: Control Group

SUMMARY:
1.Brief Introduction to the Research Background: You are invited to participate in a clinical study initiated by the First Affiliated Hospital of Zhengzhou University and chaired by Professor Zheng Yingjuan at our center. This two-year study aims to verify the sonodynamic therapy. It has been reviewed and approved for establishment by the Scientific Research Office of the First Affiliated Hospital of Zhengzhou University and has also obtained the approval of the Ethics Committee of the First Affiliated Hospital of Zhengzhou University to conduct the clinical research. This informed consent form provides you with relevant information about this clinical study to help you decide whether to participate. If you agree to participate, please read the following instructions carefully. If you have any questions, you can consult the researchers in charge of this study.

DETAILED DESCRIPTION:
2.Research Objectives (Brief Background and Significance): To evaluate the safety and efficacy of sonodynamic therapy combined with radiotherapy and chemotherapy in the treatment of brainstem gliomas, and to explore the clinical problems existing in the treatment process.

3.Research Process and Methods (Brief): Sonodynamic therapy can significantly inhibit tumor cells through mechanisms such as direct ultrasonic killing of tumor cells, generation of excessive reactive oxygen species, cavitation effects, inhibition of angiogenesis, and anti-tumor immune effects, thereby suppressing tumor growth. This trial plans to recruit 216 newly diagnosed patients with brainstem Diffuse Intrinsic Pontine Glioma (DIPG). The patients will be stratified according to factors such as their basic clinicopathological characteristics and randomly divided into an experimental group and a control group at a 1:1 ratio. Subjects in the experimental group will receive not only SDT but also treatment regimens selected by the researchers, such as radiotherapy, temozolomide, and bevacizumab. Subjects in the control group will only receive the treatment regimens selected by the researchers. The SDT treatment process is as follows: administer "Xipofen" at a dose of 5 mg/kg body weight; start sonodynamic therapy 40 minutes later; place the ultrasonic probe at the positioning point for 15 minutes, twice a day for 4 consecutive days. During the research process, we need to collect some of your specimens, which will be sampled by professionals. For example, we will collect samples for blood routine and liver and kidney function tests. Your samples will only be used for sonodynamic therapy research.

4.Potential Benefits of the Research: Detecting your specimens can help diagnose the disease, provide necessary treatment recommendations for you, or offer useful information for disease research.

5.Research Risks and Discomforts: Systemic symptoms such as phototoxic reactions, fatigue, weakness, fever, and pain; skin and mucosal symptoms such as rashes, ulcers, and bleeding; digestive tract symptoms such as diarrhea, nausea, vomiting, anorexia, and melena; respiratory system symptoms such as cough, asthma, hemoptysis, and dyspnea; as well as symptoms of the nervous and cardiovascular systems. In case of photosensitizer allergic reactions, shock, etc., the drug infusion should be stopped immediately, and anti-allergic and anti-shock treatments should be carried out.

6.Other Alternative Treatments: Chemotherapy; Radiotherapy. 7.Privacy Protection (During the Research Process and in the Publication of Results): If you decide to participate in this study, your participation in the trial and your personal data during the research will be kept confidential. All information about you will be kept confidential. For example, your blood/urine specimens will be labeled with research numbers instead of your name. Information that can identify your identity will not be disclosed to members outside the research team unless you give permission. Explain why the identifier must be retained if it is necessary. Indicate when the research materials (written or recorded in other ways) will be destroyed. If the materials are not destroyed at the end of the research, introduce where they will be stored and for how long. Explain how the stored materials will be used in the future and how to obtain the subjects' permission for future use of their materials. All research members and the research sponsor are required to keep your identity confidential. Your files will be stored in the xxx filing cabinet and only accessible to researchers. To ensure that the research is carried out in accordance with the regulations, members of the government regulatory department or the ethics review committee can review your personal data at the research unit as required if necessary. When the results of this study are published, a commitment to confidentiality is also required.

8. Voluntary Withdrawal: As a subject, you can learn about the information and progress of this research at any time and decide voluntarily whether to (continue to) participate. After participation, regardless of whether an injury occurs or how serious it is, you can choose to notify the researcher at any time to withdraw from the research. The data collected from you after withdrawal will not be included in the research results, and your medical treatment and rights will not be affected. If you continue to participate in the research and suffer serious injuries, the researcher will also stop the research. If you have questions about the research content, please contact the research doctor at ________; if you have questions related to your rights and interests, you can contact the ethics committee through the contact information at the footer of this informed consent form.

10. Sharing of Research Results after the Study: When the research is completed and the research product or intervention has been proven to be safe and effective, clarify whether it will be provided to the subjects, when and how it will be provided, and whether payment is required.

ELIGIBILITY:
Inclusion Criteria:

* 1) All subjects or their legal representatives must voluntarily and in writing sign the informed consent form approved by the ethics committee before starting the screening process;
* 2) Age < 75 years old, gender is not limited.;
* 3) Newly diagnosed patients with brainstem DIPG. It is confirmed as brainstem DIPG by histology or cytology (referring to the WHO Classification of Tumors of the Central Nervous System 2016), and there are radiologically evaluable lesions;
* 4) ECOG score is 0 - 2;
* 5) The expected survival period is ≥ 3 months;
* 6) The subjects have sufficient organ and bone marrow functions, without severe hematopoietic dysfunction and abnormal heart, lung, liver, kidney functions or immunodeficiency. The hematological indicators before enrollment are basically normal: white blood cell count ≥ 4×10⁹/L, absolute neutrophil count ≥ 1.5×10⁹/L, platelet ≥ 100×10⁹/L, hemoglobin ≥ 90 g/L. The renal function is basically normal: serum creatinine ≤ 1.2 mg/dL or creatinine clearance rate ≥ 60 ml/min. The liver function is basically normal: serum total bilirubin ≤ 1.5 × ULN (if there is liver metastasis, then serum total bilirubin should ≤ 3.0 × ULN); aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.0 × ULN (if there is liver metastasis ≤ 5.0 × ULN). The coagulation function is basically normal: the international normalized ratio of prothrombin time (INR) ≤ 2.0, and PT, APTT, and TT are all within the normal range;
* 7) The toxic reactions of anti-tumor treatment before the administration of the test drug have decreased to Grade 1 or below, or the subjects have fully recovered from previous surgeries (judged by the researcher). 8) Women of childbearing age and all male subjects must agree to use highly effective contraceptive methods during the trial period and within 12 months after the last use of hematoporphyrin injection (such as condoms, contraceptive sponges, contraceptive gels, contraceptive membranes, intrauterine devices, oral or injectable contraceptives, subcutaneous implants, etc.), and the pregnancy test results of women of childbearing age must be negative within ≤ 7 days before the administration of the test drug.

Exclusion Criteria:

* 1) Subjects known to be allergic to hematoporphyrin or other photosensitive drugs;
* 2) Subjects who participated in any other drug clinical trials or other interventional clinical trials within 4 weeks before the administration of the test drug, except for those who participated in observational (non-interventional) clinical studies or those who are in the follow-up period of interventional studies;
* 3) Subjects who have previously received SDT treatment;
* 4) Subjects who used other photosensitive drugs (tetracycline antibiotics, sulfonamides, phenothiazines, sulfonylurea hypoglycemic drugs, thiazide diuretics, and griseofulvin, etc.) within 4 weeks before the administration of the test drug
* 5) Subjects with brainstem gliomas in a cachectic state or who are expected to be unable to tolerate SDT treatment;
* 6) Subjects with uncontrolled infections or clinically significant active infectious diseases;
* 7) Subjects with positive test results for any one or more of hepatitis C virus (HCV) antibody, syphilis antibody, or human immunodeficiency virus (HIV) antibody, or subjects with active hepatitis B (defined as HBV DNA ≥ 2000 IU/mL or HBV DNA ≥ 10⁴ copies);
* 8) Difficult-to-control epilepsy and/or increased intracranial pressure and/or hypertension and/or hyperglycemia;
* 9) Subjects with severe or uncontrolled cardiovascular and cerebrovascular diseases and lung diseases (including myocardial infarction, Class III - IV heart failure, cardiac insufficiency, Grade 2 or above heart block, severe arrhythmia, cerebral infarction, cerebral hemorrhage, asthma attack, or severe respiratory failure);
* 10) Subjects who have had other malignant tumors in the past 5 years and have not been effectively controlled;
* 11) Subjects with uncontrolled mental illnesses/social situations that are expected to limit their compliance with the research requirements or impair the subject's ability to sign the informed consent form in writing;
* 12) Pregnant or lactating women;
* 13) Subjects with other reasons judged by the researcher to be unsuitable for participating in this trial, such as those with large brain tumor lesions.

Max Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2028-05-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Progression - free survival (PFS) | It is evaluated for up to 5 years from the date of randomization to the date of first documented progression or death from any cause, whichever comes first.

SECONDARY OUTCOMES:
Overall survival time | It is evaluated for up to 5 years from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- First H A Zhengzhou U, Zhengzhou, Undefined, China

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT06999148/Prot_000.pdf
  • Informed Consent Form (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT06999148/ICF_001.pdf